CLINICAL TRIAL: NCT02731066
Title: Substrate Utilization, Exercise Performance, and Skeletal Muscle Response to Energy Deficit and Altitude Acclimatization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Eastern Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-02-HC
Record Dates: First submitted 2016-03-29; First posted 2016-04-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Weight Loss; Other Effects of High Altitude
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- High pro, carbo bev (Experimental): Volunteers will receive dietary protein at 2.0 ± 0.2 g/kg/d within a 40% energy deficit diet. During aerobic performance testing, volunteers will receive a beverage containing 80 g glucose + 65 g fructose consumed at a rate providing ~1.8 g carbohydrate/min.
  Interventions: Other: High pro; Other: carbo bev
- Standard pro, carbo bev (Experimental): Volunteers will receive dietary protein at 1.0 ± 0.2 g/kg/d within a 40% energy deficit diet. During aerobic performance testing, volunteers will receive a beverage containing 80 g glucose + 65 g fructose consumed at a rate providing ~1.8 g carbohydrate/min.
  Interventions: Other: Standard pro; Other: carbo bev
- High pro, placebo bev (Experimental): Volunteers will receive dietary protein at 2.0 ± 0.2 g/kg/d within a 40% energy deficit diet. During aerobic performance testing, volunteers will receive a volume and flavor-matched, non-nutritive placebo beverage.
  Interventions: Other: High pro; Other: placebo bev
- Standard pro, placebo bev (Experimental): Volunteers will receive dietary protein at 1.0 ± 0.2 g/kg/d within a 40% energy deficit diet. During aerobic performance testing, volunteers will receive a volume and flavor-matched, non-nutritive placebo beverage.
  Interventions: Other: Standard pro; Other: placebo bev

INTERVENTIONS:
Other: Standard pro — Volunteers will receive dietary protein at 1.0 ± 0.2 g/kg/d.
  Arms: Standard pro, carbo bev; Standard pro, placebo bev
Other: High pro — Volunteers will receive dietary protein at 2.0 ± 0.2 g/kg/d.
  Arms: High pro, carbo bev; High pro, placebo bev
Other: carbo bev — During aerobic performance testing, volunteers will receive a beverage containing 80 g glucose + 65 g fructose consumed at a rate providing ~1.8 g carbohydrate/min.
  Arms: High pro, carbo bev; Standard pro, carbo bev
Other: placebo bev — During aerobic performance testing, volunteers will receive a volume and flavor-matched, non-nutritive placebo beverage.
  Arms: High pro, placebo bev; Standard pro, placebo bev

SUMMARY:
This research will evaluate nutrition requirements for missions at high altitude (i.e. >7800 feet above sea level) and the information obtained can be used to optimize nutrient content specifications for combat rations.

The objectives are:

1. Determine whether loss of lean body mass resulting from negative calorie balance over a 22-d period at high altitude can be prevented by increasing dietary protein intake.
2. Determine the efficacy of carbohydrate (glucose and fructose) supplementation on aerobic exercise performance at sea level, acute exposure to high altitude, and in response to 22-d period of negative calorie balance at high altitude.
3. Determine cognitive function, sleep patterns, and behavioral responses to high altitude and underfeeding.
4. Determine appetite and eating behavior in response to high altitude and sustained underfeeding.
5. Examine the effects of high altitude, negative calorie balance, dietary intake manipulations on gut health.

DETAILED DESCRIPTION:
Twenty-four, normal to overweight (body mass index of 18.5-29.9 kg/m2), physically active adult civilians or active duty military personnel will be recruited for the 44-d protocol, 22-d at sea level and 22-d at high altitude (HA). During the 22-d sea level phase, volunteers will receive dietary counseling to maintain baseline weight and consume protein at levels consistent with recommendations for periods of low physical activity (1.0 g/kg/d). During the 22-d at HA, all meals and beverages (water ad libitum) will be prepared and provided to volunteers by research staff. Physical activity will be increased at HA and calorie intake will be reduced 40% to create a state of negative calorie balance.

Changes in total body, lean body, and fat mass will be assessed at sea level and after a 22-d energy deficit at HA. Regulation of muscle mass will be assessed using stable isotope methodology, muscle biopsies, and various molecular techniques, to directly measure muscle protein synthesis, whole body protein balance, and the cellular mechanisms that regulate these processes. Furthermore, exercise testing, substrate oxidation rates, and expired carbon dioxide labeled with the stable isotope of carbon dioxide (one extra neutron) will be used to assess total, exogenous, and endogenous carbohydrate oxidation and performance capacity.

A comprehensive cognitive/behavioral test battery will be performed at sea level and HA. Sleep will be assessed by actigraphy. Eating behavior and appetite will be assessed at sea level, acute HA, and after the 22-d energy deficit at HA using validated measures. Gut health will be assessed using sugar absorption tests and the bacterial composition of the gut will be characterized using advanced molecular techniques.

ELIGIBILITY:
Inclusion Criteria:

* Born at altitudes less than 2,100 m (~7,000 feet)
* Physically active based on assessment of physical activity history (2-4 days per week aerobic and/or resistance exercise)
* Body weight ≥ 110 lbs.
* Body mass index (BMI) between 18.5-29.9 kg/m2
* Females must be on contraception (e.g., oral birth control, NuvaRing®, Depo Provera®, etc.)
* Have supervisor approval (permanent party military)
* Not taking any medications and/or willing to refrain from all medication use 4 wk prior to and throughout the entire study period, unless provided/approved by the US Army Research Institute of Environmental Medicine (USARIEM) Office of Medical Support and Oversight (OMSO) or medical oversight at Pikes Peak, Colorado organized through OMSO.
* Willing to refrain from alcohol, smoking any nicotine product (includes e-cigarettes), electronic cigarettes, chewing tobacco, caffeine, and dietary supplement use throughout the entire study period
* Willing to travel to USARIEM's Altitude Laboratory at Pikes Peak and live there for 22 consecutive days
* Refrain from taking any nonsteroidal anti-inflammatory drugs (NSAIDs; e.g. aspirin, Advil®, Aleve®, Naprosyn®, or any aspirin-containing product) for 10 days before and at least 5 days AFTER each muscle biopsy. (*Tylenol® or acetaminophen is ok to use if needed for discomfort)

Exclusion Criteria:

* Born at altitudes greater than 2,100 m (~7,000 feet)
* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for five days or more within the last 2 mo
* Musculoskeletal injuries that compromise exercise capability
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Disease or medication that affects macronutrient metabolism and/or the ability to participate in strenuous exercise
* Evidence of apnea or other sleeping disorders
* Evidence of prior high altitude pulmonary edema or high altitude cerebral edema diagnosis
* Allergies or intolerance to foods (including but not limited to lactose intolerance/milk allergy), vegetarian practices, or medications (including, but not limited to, lidocaine or phenylalanine) to be utilized in the study
* History of complications with lidocaine
* Taking medications that interfere with oxygen delivery and transport (Includes sedatives, sleeping aids, tranquilizers and/or any medication that depresses ventilation, diuretics, alpha and beta blockers)
* Evidence of any physical, mental, and/or medical conditions that would make the proposed studies relatively more hazardous as determined by OMSO
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Anemia (hematocrit <38% for males, <36% for females, and hemoglobin >12.5 g/dL for all subjects) or Sickle Cell Anemia/Trait
* Abnormal prothrombin time/partial thromboplastin time (PT/PTT) test or problems with blood clotting
* Blood donation within 8 weeks of beginning the study
* Pregnancy and women not on contraceptives
* Any use of antibiotics, except topical antibiotics, within 3 months of study participation.
* Colonoscopy within 3 months of study participation
* Use of laxatives, stool softeners, or anti-diarrheal medications at least once a week.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in lean body mass | baseline (sea level day 0), prior to altitude exposure (sea level day 20), after ~3 wk energy deficit diet at high altitude (high altitude day 19)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Pasiakos, PhD, Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Berryman CE, Young AJ, Karl JP, Kenefick RW, Margolis LM, Cole RE, Carbone JW, Lieberman HR, Kim IY, Ferrando AA, Pasiakos SM. Severe negative energy balance during 21 d at high altitude decreases fat-free mass regardless of dietary protein intake: a randomized controlled trial. FASEB J. 2018 Feb;32(2):894-905. doi: 10.1096/fj.201700915R. Epub 2018 Jan 3. PMID 29066613
- [Derived] Hennigar SR, Berryman CE, Kelley AM, Anderson BJ, Young AJ, McClung JP, Pasiakos SM. High-Altitude Acclimatization Suppresses Hepcidin Expression During Severe Energy Deficit. High Alt Med Biol. 2020 Sep;21(3):232-236. doi: 10.1089/ham.2019.0109. Epub 2020 Apr 21. PMID 32316799
- [Derived] Bradbury KE, Berryman CE, Wilson MA, Luippold AJ, Kenefick RW, Young AJ, Pasiakos SM. Effects of carbohydrate supplementation on aerobic exercise performance during acute high altitude exposure and after 22 days of acclimatization and energy deficit. J Int Soc Sports Nutr. 2020 Jan 9;17(1):4. doi: 10.1186/s12970-020-0335-2. PMID 31918720